CLINICAL TRIAL: NCT07028229
Title: Development and Validation of an Ultrasound Training Program for Residents in Staging Gynecological Cancers (Ovarian Cancer, Endometrial Cancer and Cervical Cancer)
Brief Title: Ultrasound Training Program for Gynecologic Cancer Staging in Residents
Acronym: Ultra-teaching
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7738
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Medical Education; Ovarian Cancer; Endometrial Cancer; Cervix Cancer
Keywords: Resident Training; Learning Curve; Gynecologic Oncology; Transvaginal Ultrasound
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Experimental): Gynecology and obstetrics residents enrolled in a structured ultrasound training program focused on staging of gynecologic cancers. The program includes theoretical lessons, supervised hands-on sessions, and independent ultrasound assessments compared with expert findings.
  Interventions: Behavioral: Training Group

INTERVENTIONS:
Behavioral: Training Group — A structured educational and practical training program in gynecologic oncology ultrasound designed for residents. The intervention includes lectures, clinical case discussions, supervised and independent ultrasound examinations, and performance assessments to evaluate learning progression and diagnostic concordance with experts.
  Other Names: Ultrasound Training Program for Gynecologic Cancer Staging

SUMMARY:
This is a prospective, interventional study aiming to develop and validate an ultrasound training program for gynecology and obstetrics residents, focused on the staging of gynecologic cancers, including ovarian, endometrial, and cervical cancer. The program consists of theoretical lectures, practical hands-on sessions, and supervised clinical case evaluations over a six-month period. Residents will perform ultrasound examinations independently, which will be compared to those conducted by expert sonographers. The primary objective is to assess the learning curve of each trainee by evaluating diagnostic concordance with expert findings across specific staging parameters.

ELIGIBILITY:
Inclusion Criteria:

* At least six gynecology residents who will regularly attend the ultrasound center daily, with overlapping shifts.
* All patients with a diagnosis or suspected diagnosis of gynecological cancer, including ovarian, endometrial, and cervical cancers, will be included in the study and scanned by both residents and experts.
* Signing of the informed consent by the participants.

Exclusion Criteria:

* non-gynecology specialists, with attendance schedules at the center other than daily.
* Failure to sign the informed consent by the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study enrolls female patients diagnosed or suspected of having gynecologic cancers (ovarian, endometrial, or cervical cancer) who undergo ultrasound examinations. Medical residents of any gender specializing in gynecology and obstetrics are eligible to participate as trainees in the ultrasound training program.
Enrollment: 6 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Agreement Rate Between Residents and Experts in Ultrasound-Based Staging of Gynecologic Cancers | Up to 6 months (from the start to the end of the training program)
  Assessment of the diagnostic concordance between ultrasound staging performed by residents and expert sonographers, measured across defined anatomical and pathological parameters (e.g., lymph node involvement, carcinomatosis, tumor size and spread). Concordance will be quantified as the percentage of agreement per case and per parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Carla Testa, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy